CLINICAL TRIAL: NCT01368471
Title: MASTER: MGUARD for Acute ST Elevation Reperfusion
Brief Title: Safety and Efficacy Study of MGuard Stent After a Heart Attack
Acronym: MASTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: InspireMD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMD-07
Record Dates: First submitted 2011-02-17; First posted 2011-06-08 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Myocardial Infarction
Keywords: STEMI; myocardial infarction; stent
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MGuard (Experimental): MGuard stent will be deployed
  Interventions: Device: MGuard
- BMS or DES (Active Comparator): A regular bare metal stent or drug-eluting stent will be deployed
  Interventions: Device: Control BMS or DES

INTERVENTIONS:
Device: MGuard — MGuard™ stent comprises a balloon-expandable, thin-strut stainless steel (316L) bare metal stent platform (strut width 100 µm) with mesh sleeve fibers of polyethyleneterephtalate (fiber width of 20 µm) attached to its outer surface. These fibers act like a net (aperture size 150 x 180 µm) preventing distal embolization of the plaque debris/thrombus placed between the vessel wall and the stent.
  Arms: MGuard
Device: Control BMS or DES — Control BMS or DES
  Arms: BMS or DES

SUMMARY:
The goal of this study is to demonstrate the superiority of the MGuard™ stent over commercially-approved bare-metal (BMS) /drug-eluting stents (DES) in achieving better myocardial reperfusion in primary angioplasty for the treatment of acute ST-elevation myocardial infarction (STEMI).

ELIGIBILITY:
Inclusion Criteria

* 18 years of age
* ST-segment elevation (more than 2mm in more than contiguous leads)
* MI with symptom onset less than 12h
* The patient is willing to comply with specified follow-up evaluations
* Signed ICF
* Single de novo lesion in the target (culprit) vessel
* Target lesion maximum length is 33 mm (by visual estimation)
* Reference vessel diameter must be more than 3.0 to less than 4.0 mm by visual estimation
* Randomization should occur as soon as Presence of TIMI 2 or 3 before randomization Exclusion Criteria
* Pregnant or nursing patients
* Left Bundle Branch Block (LBBB), paced rhythm, or other Electrocardiogram (ECG) abnormality
* Impaired renal function
* Prior coronary artery bypass graft surgery
* Bleeding diathesis
* Contraindication to aspirin
* cardiopulmonary resuscitation
* Cardiogenic shock
* chronic warfarin anticoagulation
* LVEF less than 20%
* other medical illness
* participation in another investigational drug or device study that has not reached its primary endpoint
* Left main coronary artery disease with 50% stenosis
* Ostial target lesion
* Failure to visualize vessel anatomy distal to the culprit lesion
* Moderate to heavily calcified target lesion or vessel
* excessive tortuosity
* bifurcation with a side branch more than 2.0 mm in diameter
* A significant (greater than 50%) stenosis proximal or distal to the target lesion is present that cannot be covered by same single stent
* Diffuse disease distal to target lesion with impaired runoff
* Any prior stent proximal to the target lesion, or within 10 mm distal of the target lesion
* PCI of another lesion performed within 6 months before the index procedure
* Target lesion located in a saphenous vein graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The incidence of complete ST segment resolution (defined as ≥70% ST 1. The incidence of complete ST segment resolution | 60 to 90 minutes after the last angiogram

SECONDARY OUTCOMES:
The incidence of Thrombolysis In Myocardial Infarction (TIMI) 3 flow at the end of the procedure. | 60-90 minutes after last angiogram
  The incidence of TIMI 3 flow at the end of the procedure.
Major Adverse Cardiac Events (MACE)at discharge, 30 days, 6 months and 12 months post-procedure | discharge, 30 days, 6 and 12 months post-procedure
  Major Adverse Cardiac Events (MACE): defined as cardiac death, reinfarction (Q wave and non-Q wave), or repeat ischemia-driven target lesion revascularization (TLR) by percutaneous or surgical methods at hospital discharge, 30 days, 6 months and 1 year post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Abizaid, MD, PhD, Principal Investigator — Inst Dante Pazzanese of Cardiology, Brazil; Dariusz Dudek, MD, PhD, Principal Investigator — Cardiac Catheterization Laboratories, Krakow, Poland; Sigmund Silber, MD, PhD, Principal Investigator — Heart Center at the Isar Academic Teaching Site of the University of Munich; Gregg Stone, MD, Study Chair — Columbia University Medical Center The Cardiovascular Research Foundation
Locations (7):
- Poland (6):
  - Klinika Kardiologii Inwazyjnej Uniwersytetu Medycznego w Białymstoku, Bialystok
  - Gilghsin: John Paul II Hospital, Krakow
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Oddział Kardiologii Inwazyjnej, Nowy Targ
  - Centrum Kardiologii Inwazyjnej GVM Carint, Oświęcim
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
- Milpark Hospital, Johannesburg, South Africa

REFERENCES:
- [Derived] Dudek D, Dziewierz A, Brener SJ, Abizaid A, Merkely B, Costa RA, Bar E, Rakowski T, Kornowski R, Dressler O, Abizaid A, Silber S, Stone GW. Mesh-covered embolic protection stent implantation in ST-segment-elevation myocardial infarction: final 1-year clinical and angiographic results from the MGUARD for acute ST elevation reperfusion trial. Circ Cardiovasc Interv. 2015 Feb;8(2):e001484. doi: 10.1161/CIRCINTERVENTIONS.114.001484. PMID 25603802
- [Derived] Dudek D, Brener SJ, Rakowski T, Dziewierz A, Abizaid A, Silber S, Yaacoby E, Dizon JM, Costa RA, Maehara A, Dressler O, Stone GW. Efficacy of an Embolic Protection Stent as a Function of Delay to Reperfusion in ST-Segment Elevation Myocardial Infarction (from the MASTER Trial). Am J Cardiol. 2014 Nov 15;114(10):1485-9. doi: 10.1016/j.amjcard.2014.08.007. Epub 2014 Aug 27. PMID 25277335
- [Derived] Stone GW, Abizaid A, Silber S, Dizon JM, Merkely B, Costa RA, Kornowski R, Abizaid A, Wojdyla R, Maehara A, Dressler O, Brener SJ, Bar E, Dudek D. Prospective, Randomized, Multicenter Evaluation of a Polyethylene Terephthalate Micronet Mesh-Covered Stent (MGuard) in ST-Segment Elevation Myocardial Infarction: The MASTER Trial. J Am Coll Cardiol. 2012 Nov 6;60(19):1975-84. doi: 10.1016/j.jacc.2012.09.004. PMID 23103033